CLINICAL TRIAL: NCT03257657
Title: Helping Moms to be Healthy After Baby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-1932; UL1TR002535 (NIH)
Record Dates: First submitted 2017-08-01; First posted 2017-08-22 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Weight Loss; Diet Modification; Obesity
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: This is a pilot, randomized controlled trial. The investigators will pilot a multi-component intervention delivered in a WIC (Women, Infants, children) setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational Group (Experimental): Intervention: Participants will receive usual WIC care plus they will be given a packet of written WIC materials on lifestyle recommendations at the baseline visit, and offered an appointment with a WIC Registered Dietitian (RD) at the 12 week visit.
  Interventions: Behavioral: Observation Group participants
- Lifestyle Group (Experimental): Intervention: Visits with WIC staff at Baseline, 4 weeks, 8 weeks: Meet with WIC staff who will use motivational interviewing during visits. Participants will complete an iPad app that asks lifestyle questions. Responses are provided to WIC staff in an easy to read format to guide lifestyle counseling and informational handouts are provided to participants.
  In-between visits: Participants receive text messages with informational and motivational content. They are invited to a Facebook private group providing informational and motivational content and encouraging cross-support amongst participants. They are asked to self-monitor activity and weekly weights and will be offered weekly phone coaching appointments with WIC staff.
  Interventions: Behavioral: Lifestyle group participants

INTERVENTIONS:
Behavioral: Observation Group participants — Women in the observation group will receive usual WIC care, plus the opportunity to meet with a WIC Registered Dietitian (RD) at the 12 week visit. Written WIC materials on lifestyle recommendations will also be given to all observation group participants at the baseline visit. The Investigators will connect with the participant prior to the 12 week visit to make an appointment to meet with the WIC RD at that time.
  Arms: Observational Group
Behavioral: Lifestyle group participants — Women in this group will receive typical WIC care plus the below described activities. The intervention will last 12 weeks.
  Arms: Lifestyle Group

SUMMARY:
Low-income and minority women are at increased risk for postpartum weight retention (i.e. retaining weight after pregnancy) and consequent persistent obesity. Women who are obese pre-pregnancy are 3-5 times more likely to gain weight, rather than lose weight, in the postpartum period than non-obese women. Aims for this pilot study are listed below:

Aim 1: To evaluate the feasibility and acceptability of a multi-component novel weight loss intervention delivered in a WIC setting to a population of low-income, predominantly racial/ethnic minority, obese, postpartum women.

Aim 2: To evaluate differences in weight change, diet, physical activity, self-efficacy, readiness to change, motivations to eat between intervention and control participants to determine preliminary intervention efficacy over a 12-week period.

DETAILED DESCRIPTION:
Low-income and minority women are at increased risk for postpartum weight retention (i.e. retaining weight after pregnancy) and consequent persistent obesity. Women who are obese pre-pregnancy are 3-5 times more likely to gain weight, rather than lose weight, in the postpartum period than non-obese women.

Obesity science supports that weight loss interventions should be multi-component with regular points of contact. Building upon this, we have designed a multi-component intervention that considers the demands on women in the postpartum period and utilizes technology for both provider decision support and for virtual contact with participants. The intervention will address diet, physical activity, and social support through the use of in-person meetings with WIC staff, text messaging, phone coaching, self-monitoring, and Facebook.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥18 and <50 years old).
* Enrolled in WIC or with an infant enrolled in WIC.
* 3-12 months postpartum.
* A pre-pregnancy BMI of 25 - 40 kg/m2 (based on self-reported height and weight prior to pregnancy).
* Postpartum body mass index between 25 and 50 kg/m2.
* English- and/or Spanish-speaking.
* Owns a mobile phone with texting functionality in order to receive texts during the trial.

Exclusion Criteria:

* Health conditions impacting weight or ability to participate in a weight loss trial.
* Pregnancy or planned pregnancy in next 5 months.
* Any health problems or undergoing any treatments that might interfere with what participant eats or her ability to exercise.
* Medical provider recommendation to avoid exercise.
* Plans to be in a different geographic area within the next 5 months.
* Plans to stop coming to Aurora WIC in the next 5 months.
* Unable to give informed consent.
* Not able to read and understand English or Spanish at an 8th grade level.
* Not willing to create a Facebook account if they do not already have one.
* Asked to follow-up in < 3 months at most recent WIC visit.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darcy A Thompson, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Aurora WIC Office, Aurora, Colorado
  - University of Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lifestyle Group: Intervention: Visits with WIC staff at Baseline, 4 weeks, 8 weeks: Meet with WIC staff who will use motivational interviewing during visits. Participants will complete an iPad app that asks lifestyle questions. Responses are provided to WIC staff in an easy to read format to guide lifestyle counseling and informational handouts are provided to participants.
  In-between visits: Participants receive text messages with informational and motivational content. They are invited to a Facebook private group providing informational and motivational content and encouraging cross-support amongst participants. They are asked to self-monitor activity and weekly weights and will be offered weekly phone coaching appointments with WIC staff.
  Lifestyle group participants: Women in this group will receive typical WIC care plus the below described activities. The intervention will last 12 weeks.
Period: Overall Study
Arm/Group | Observational Group | Lifestyle Group
Started | 22 | 20
Completed | 22 | 15
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawn | 0 | 1
Not completed — Noted not eligible right after enrolled | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observational Group | Lifestyle Group | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (6.6) | 30.5 (5.0) | 30.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 20 | 17 | 37
  African American, non-Hispanic | 1 | 2 | 3
  White, non-Hispanic | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment
Description: The investigators plan to determine the feasibility of recruitment for a weight loss intervention by evaluating the rate of recruitment. Below describes number recruited/enrolled over 14 weeks of recruitment
Time Frame: Once the final participant is recruited
Population: One participant was consented but determined before receiving any interventions that they did not meet all eligibility criteria. This participant is excluded from the lifestyle group.
Measure: Number; unit: participants
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 19
participants | 22 | 19

2. Primary Outcome: Attrition Rate of Subjects Enrolled in the Study
Description: The investigators will measure the number of dropouts/withdrawn once final participant has completed the 12 week visit.
Time Frame: Once the final participant completes the 12 week visit
Population: The 1 participant originally enrolled, but removed right after enrollment because was determined not eligible is not included in the Lifestyle group count.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 19
Participants | 0 | 4

3. Primary Outcome: Visit Attendance
Description: The investigators will measure lifestyle group participant attendance from enrollment through the 12-week visit. The number of participants who attended their visits is reported
Time Frame: Baseline through Week 12, reported at Week 12
Population: 2 participants are excluded from analysis: Participant who was withdrawn was not included in analysis. Participant identified as not eligible right after enrollment is not included either.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Group
Number analyzed (Participants) | 18
Participants
  Attended all 4 visits (Baseline, 4 week visit, 8 | 7
  Attended 3 of 4 visits (Baseline, 4 or 8 week visi | 5
  Attended 2 of 4 visits (baseline and 12 week visi | 3
  Attended 0 intervention visits | 3

4. Primary Outcome: Acceptability of a Weight Loss Intervention
Description: To determine acceptability, investigators will use qualitative interviews to ask open-ended questions on this topic including asking participants in the intervention whether they would participate again. The number of participants interviewed who indicated that they would participate again is reported.
Time Frame: 12 weeks
Population: Data was not available for analysis for one participant. This participant was not analyzed. The three participants lost to follow-up before the baseline visit were not available for interview and are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle Group
Number analyzed (Participants) | 14
Participants | 14

5. Primary Outcome: Evaluation of the Use of Phone Coaching
Description: Investigators will count the total number of times any participant used phone coaching.
Time Frame: 12 weeks
Measure: Number; unit: Number of phone coaching sessions
Arm/Group | Lifestyle Group
Number analyzed (Participants) | 19
Number of phone coaching sessions | 1

6. Secondary Outcome: Change in Weight Between Visits
Description: To determine differences in change in weight between the intervention and control groups, participants will be weighed on a scale in the Women, Infants, and Children (WIC) setting.
Time Frame: Intervention group: Baseline, 12 weeks; Control group: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 15
pounds | -0.8 (6.4) | -4.7 (7.5)
Statistical Analysis 1: Comparison: Observational Group vs Lifestyle Group; Test type: Other; p = 0.1, t-test, 2 sided

7. Secondary Outcome: Changes in Diet: Intakes Measured in Grams
Description: To determine differences in diet from baseline to 12 weeks between intervention and control groups, participants will complete the Block Fat-Sugar-Fruit-Vegetable Screener. This is a validated food screener for adults.
Time Frame: Baseline and 12 weeks
Population: Data missing for one Lifestyle Group participant at the 12 week point
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 14
Grams
  Saturated fat (g) | -3.7 (8.1) | -4.1 (5.7)
  Trans fat (g) | 0.2 (3.5) | -1.2 (2.7)
  Total sugars (g) | -35.1 (50.4) | -25.2 (34)
  Added sugars (g) | -25.7 (39.5) | -23.3 (33.6)
  protein (g) | -10.2 (22.2) | -6.3 (25.5)
  total fat (g) | -9.9 (24.5) | -9.4 (16.4)
  carbohydrates (g) | -40.9 (79.8) | -46.7 (48.8)
  fiber (g) | 0.1 (4.8) | -0.4 (3.1)

8. Secondary Outcome: Changes in Physical Activity
Description: To determine differences in total physical activity from baseline to 12 weeks between intervention and control groups, participants will complete an adapted version of the Pregnancy Physical Activity Questionnaire. This is a validated survey measure for physical activity.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: MET-h/week
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 15
MET-h/week | -45.5 (176) | 38.6 (126)
Statistical Analysis 1: Comparison: Observational Group vs Lifestyle Group; Test type: Other; p = 0.13, t-test, 2 sided

9. Secondary Outcome: Changes in Diet and Physical Activity Self-efficacy
Description: To determine differences in self-efficacy from baseline to 12 weeks between intervention and control groups, participants will complete an adapted version of Eating Habits Confidence Survey and Exercise Confidence Survey.
  Diet self-efficacy: Possible range: -32 to 32; Higher scores indicate improved self-efficacy.
  Physical activity self-efficacy: Sticking to it scale: Possible range: -32 to 32; Higher scores indicate improved self-efficacy.
  Making time scale: -12 to 12; Higher scores indicate improved self-efficacy.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 14
units on a scale
  Physical activity: Sticking to it | -0.5 (0.9) | 0.4 (1.0)
  Physical activity: making time for exercise | -0.3 (1.0) | 0.0 (0.8)
  Diet | 3.3 (3.1) | -0.1 (7.2)

10. Secondary Outcome: Changes in Motivations to Eat
Description: To determine differences from baseline to12 weeks in motivations to eat between intervention and control groups, participants will complete the Eating Stimulus Index questionnaire.
  Possible range = -92 to 92. Higher scores indicated improved lifestyle-related behaviors and motivations to eat.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 14
units on a scale | -3.3 (9.6) | 5.9 (12.0)
Statistical Analysis 1: Comparison: Observational Group vs Lifestyle Group; Test type: Other; p = 0.02, t-test, 2 sided

11. Secondary Outcome: Changes in Readiness to Change
Description: Investigators will evaluate any differences in readiness to change from baseline to 12 weeks between intervention and control groups by participants completing the Readiness to Change questionnaire. Possible range = -3 to 3; higher scores indicate greater change in readiness to change
Time Frame: Baseline and 12 weeks
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 14
units on a scale
  Losing weight | 0 [0 to 1] | 1.0 [0 to 1]
  Healthy eating | 0 [0 to 1] | 1.0 [0 to 1]
  Physical activity | 0 [-1 to 1] | 1.0 [0 to 2]

12. Secondary Outcome: Changes in Diet: Intakes Measured in Cups
Description: To determine differences in diet from baseline to 12 weeks between intervention and control groups, participants will complete the Block Fat-Sugar-Fruit-Vegetable Screener. This is a validated food screener for adults. Fruit and vegetable intake changes are measured and reported in cups.
Time Frame: Baseline and 12 weeks
Population: Data missing for one Lifestyle Group participant at the 12 week point
Measure: Mean (Standard Deviation); unit: Cups
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 14
Cups
  Fruit and fruit juice (cups) | -0.2 (1.5) | 0 (1.4)
  vegetable intake (cups) | -0.1 (0.9) | 0.3 (0.9)

13. Secondary Outcome: Changes in Diet: kCal Intake
Description: as for outcome 7
Time Frame: Baseline and 12 weeks
Population: Data missing for one Lifestyle Group participant at the 12 week point
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Observational Group | Lifestyle Group
Number analyzed (Participants) | 22 | 14
kcal | -294 (531.7) | -297 (374.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Observational Group | Lifestyle Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03257657/Prot_SAP_000.pdf